CLINICAL TRIAL: NCT06362460
Title: Single-center, Open-label, Non-randomized and Single-dose Clinical Trial to Explore the Mass Balance of Oral Suspension of 400mg [14C]RAY1216
Brief Title: Mass Balance Study of [14C]RAY1216 in Healthy Adult Male Subjects in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RAY1216-23-03
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]RAY1216 (Experimental)
  Interventions: Drug: [14C] RAY1216

INTERVENTIONS:
Drug: [14C] RAY1216 — 400 mg suspension containing 100μCi of [14C]RAY1216

SUMMARY:
This study is a single-center, open-label, and single-dose clinical study to evaluate the mass balance, biotransformation and pharmacokinetics of [14C]RAY1216 in healthy Chinese male participants, revealing the overall pharmacokinetic characteristics of RAY1216.

ELIGIBILITY:
Inclusion Criteria:

1. Males and female participants between 18-45 years (Both inclusive);
2. Body weight≥50kg.Body mass index (BMI) 18~28 kg/m2 (Both inclusive); BMI is determined by the following equation: BMI = weight/height2 (kg/m2);
3. Participants who voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions.

Exclusion Criteria:

1. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests. History or presence of a clinically significant gastrointestinal, renal, hepatic, neurologic, hematic, endocrine, neoplastic, pulmonary, immune, psychiatric or cardiovascular and cerebrovascular disorder(s) (but not limited to above disorders).
2. Presence of human immunodeficiency virus (HIV), viral hepatitis(including hepatitis C virus (HCV) or hepatitis B virus (HBV) ,treponema pallidum antibodies at screening.
3. Participants who donated blood or bleeding profusely(> 400 mL)in the 3 months preceding study screening.
4. Participants who have undergone surgery within 6 months before the screening period or whose surgical incision is not completely healed; Major surgery includes, but is not limited to, any surgery with a significant risk of bleeding, or an open biopsy or significant traumatic injury;
5. Workers engaged in conditions requiring long-term exposure to radioactivity; Or have significant radiation exposure (≥2 chest/abdomen CT, or ≥3 other types of X-ray examinations) within 1 year before this study or have participated in the radiopharmaceutical labeling test;
6. Participants who smoked an average of >5 cigarettes per day in the previous 3 months or habitually used nicotine-containing products and were unable to quit during the trial period;
7. Substance abuse or use of soft drugs (e.g., marijuana) in the 3 months prior to the screening period or use of hard drugs (e.g., cocaine, amphetamines, etc.) in the 1 year prior to the screening period; Or screening for positive urine drug abuse (drug) tests;
8. Participants who have special dietary requirements and cannot comply with a uniform diet;
9. History of allergic conditions or allergic diseases, or a history of allergic reactions attributed to RAY1216 or any of the ingredients of its formulation or similar drugs.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in plasma PK | Up to 7 days from the start of administration.
  Cmax
Total radioactivity in plasma PK | Up to 7 days from the start of administration.
  AUC0-t
Total radioactivity in plasma PK | Up to 7 days from the start of administration.
  CL/F
Total radioactivity in plasma PK | Up to 7 days from the start of administration.
  Vz/F
Mass balance recovery of total radioactivity in all (urine, faeces) amount excreted (Ae) expressed as a percentage of the administered dose (%Ae) | Up to 14 days from the start of administration.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Up to 14 days (approx) from the start of administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, China